CLINICAL TRIAL: NCT00185250
Title: Double-Blind, Placebo-Controlled, Randomized, Parallel Group, Multicenter Study to Evaluate Efficacy and Safety of 4 and 8 Million Units Betaferon®/Betaseron® (Interferon Beta-1b) Given Subcutaneously Every Other Day Over 24 Weeks in Patients With Chronic Viral Cardiomyopathy
Brief Title: Betaferon/ Betaseron (Interferon Beta-1b) in Patients With Chronic Viral Cardiomyopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Schering Pharma AG
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 91115; 305852
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2008-12-19 (Estimated); Status verified 2008-12

CONDITIONS: Cardiomyopathies; Heart Diseases
Keywords: Cardiomyopathy; idiopathic chronic heart failure; Adenovirus; Enterovirus; Parvovirus
MeSH Terms: conditions — Cardiomyopathies; Heart Diseases; Adenoviridae Infections; Enterovirus Infections; Parvoviridae Infections | interventions — Interferon beta-1b

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1 (Experimental)
  Interventions: Drug: Interferon beta-1b (Betaferon/Betaseron, BAY86-5046)
- Arm 2 (Experimental)
  Interventions: Drug: Interferon beta-1b (Betaferon/Betaseron, BAY86-5046)
- Arm 3 (Placebo Comparator)
  Interventions: Drug: Placebo
- Arm 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Interferon beta-1b (Betaferon/Betaseron, BAY86-5046) — 2 MIU per application in week 1 and 4 MIU per application in weeks 2 to 24 given subcutaneously every other day
  Arms: Arm 1
Drug: Interferon beta-1b (Betaferon/Betaseron, BAY86-5046) — 2 MIU per application in week 1, 4 MIU per application in weeks 2 to 3 and 8 MIU per application in weeks 4 to 24 given subcutaneously every other day
  Arms: Arm 2
Drug: Placebo — 0.25 ml in week 1 and 0.50 ml in weeks 2 to 24 given subcutaneously every other day
  Arms: Arm 3
Drug: Placebo — 0.25 ml in week 1, 0.50 ml in weeks 2 to 3 and 1.00 ml in weeks 4 to 24 given subcutaneously every other day
  Arms: Arm 4

SUMMARY:
Chronic viral cardiomyopathy is a disease where the cardiac muscle is attacked by a virus and this may result in a reduction in the output of the heart (pump function) thereby causing complaints such as chest pain, shortness of breath and palpitations.

Betaferon (interferon beta-1b) is marketed for the treatment of Multiple Sclerosis already, but until now, it has not been proven whether it is also effective in patients with chronic viral myocardial disease.

This study will be conducted to examine the efficacy and safety of Betaferon in patients with this disease. The aim of the treatment is to eliminate the virus from the heart so that the heart function and clinical status can gradually improve.

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.

Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Unexplained heart with evidence of Adeno-, Entero- and/or Parvoviruses which must be identified directly in the heart tissue
* Being in a chronic (at least 6 month after the onset of clinical symptoms) and stable phase of the disease
* Impaired cardiac function

Exclusion Criteria:

* Severe (decompensated) or acute heart failure.
* Any other disease which could better explain the patient's clinical symptoms
* Any other severe and/or malignant disease.
* Suffering from convulsions, depression or suicidal ideas judged by a physician
* Serious viral or bacterial infections during the last weeks
* Pregnancy or lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2002-12; Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Presence of Adenovirus, Enterovirus and/or Parvovirus in endomyocardium | 12 weeks after the end of a 24 weeks treatment

SECONDARY OUTCOMES:
Changes in NYHA functional class | 12 weeks and 24 weeks after the end of treatment
Six-minute walking test | 12 weeks and 24 weeks after the end of treatment
Single clinical symptoms (dyspnea, fatigue, palpitation, atypical angina and angina pectoris) | 12 weeks and 24 weeks after the end of treatment
Quality of life | 12 weeks and 24 weeks after the end of treatment
Left ventricular ejection fraction at rest and on exertion | 12 weeks after the end of treatment
Regional and global wall motion, left ventricular enddiastolic diameter, and left ventricular endsystolic diameter | 12 weeks after the end of treatment
Inflammatory state in endomyocardial biopsies | 12 weeks after the end of treatment
Peripheral blood analyses for viral treatment effect and disease markers | 12 weeks after the end of treatment
Composite clinical endpoint | 12 weeks and 24 weeks after the end of treatment
Hemodynamics | 12 weeks after the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (30):
- France (2):
  - Nantes
  - Poitiers
- Germany (21):
  - Bad Krozingen, Baden-Wurttemberg
  - Ulm, Baden-Wurttemberg
  - München, Bavaria
  - Brandenburg, Brandenburg
  - Hamburg, Hamburg
  - Göttingen, Lower Saxony
  - Greifswald, Mecklenburg-Vorpommern
  - Rostock, Mecklenburg-Vorpommern
  - Bad Oeynhausen, North Rhine-Westphalia
  - Cologne, North Rhine-Westphalia
  - Dortmund, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Münster, North Rhine-Westphalia
  - Wuppertal, North Rhine-Westphalia
  - Ludwigshafen am Rhein, Rhineland-Palatinate
  - Homburg, Saarland
  - Leipzig, Saxony
  - Halle, Saxony-Anhalt
  - Kiel, Schleswig-Holstein
  - Berlin, State of Berlin
  - Bad Berka, Thuringia
- Italy (3):
  - Bergamo, BG
  - Milan, MI
  - Pavia
- Warsaw, Poland
- Madrid, Madrid, Spain
- Gothenburg, Sweden
- Glasgow, United Kingdom